CLINICAL TRIAL: NCT04732507
Title: Investigating the Minimum Number of Needling Required to Optimize Trigger Point Injections Outcome
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Mohab Ibrahim, PhD MD, Professor, Anesthesiology, University of Arizona
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 04122020
Record Dates: First submitted 2020-12-10; First posted 2021-02-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Myofascial Pain; Myofascial Trigger Point Pain
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Depending on assignment, one group will receive 1-2 needle passes at each trigger point, the other will receive 10 and the third will receive 20.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- One to two needle passes (Active Comparator): Receive 1-2 needle passes for needling at each trigger point
  Interventions: Combination Product: 1% plain lidocaine and 0.25% plain bupivacaine
- Ten needle passes (Active Comparator): Receive 10 needle passes for needling at each trigger point
  Interventions: Combination Product: 1% plain lidocaine and 0.25% plain bupivacaine
- Twenty needle passes (Active Comparator): Receive 20 needle passes for needling at each trigger point
  Interventions: Combination Product: 1% plain lidocaine and 0.25% plain bupivacaine

INTERVENTIONS:
Combination Product: 1% plain lidocaine and 0.25% plain bupivacaine — A 5- or 10-ml syringe will be filled equally with 1% plain lidocaine and 0.25% plain bupivacaine. A 1.5-inch 25-gauge needle will be attached to the syringe. The needle will be carefully inserted at the first trigger point and 2 mls of the mixed local anesthetic will be infiltrated. At that point, the needle will be carefully inserted into the trigger point based on the group assigned. Once needling is done for the first trigger point, the process will be repeated in exactly the same fashion for the remaining points.

SUMMARY:
Myofascial pain is a common condition in which patients may experience severe chronic pain. The source of this pain is typically the soft tissue. Current methods to address myofascial pain include a procedure called Trigger point Injections. This method involves identifying the areas of muscles that are causing the pain. The most common way to perform trigger point injection involves infiltrating the muscle with local anesthetics and then repeatedly passing the numbing needle in and out of the muscles (needling). This procedure is successful for most patients. However, there is great variability in the way needling is done. Some pain physicians perform 1-2 needle passes while other pain physicians may exceed 20 passes. There are currently no guidelines as to the number or amount of needle passes needed to achieve pain control. Furthermore, there is no study or research to shed light on the relationship between the number of needles passes and the degree and duration of pain relief coupled with patients' satisfaction.

This study is proposed to address this gap in knowledge. It is a prospective and randomized clinical trial that follows the standard of care. The investigators will recruit patients from The University-Banner Medical Center at Tucson, Arizona chronic pain clinic who are candidates for trigger point injections. The participants will be randomized into 3 different groups. Group one will receive 2 needle passes per identified trigger point. Group two will receive ten needle passes per identified trigger point. Group three will receive twenty needle passes per identified trigger point.

The investigators will analyze the data to understand the relationship between the number of needles passes and the degree of pain relief, improved functional capacity, and patients' satisfaction.

DETAILED DESCRIPTION:
Chronic pain affects over 100 million Americans with an annual cost of about $600 billion/year. Almost half of the chronic pain conditions are attributed to musculoskeletal conditions.

Musculoskeletal pain is typically identified with palpation over tender areas initially identified by the patient and then verified by the physician. There are typically areas of muscles that when palpated, pain is experienced by the patient. These points are known as Trigger Points. There are several ways to manage trigger points. Muscle relaxers are the most common pharmacological approaches to manage trigger points, but they can cause significant sedation for patients. Some non-pharmacological methods such as physical therapy may also provide some relief of musculoskeletal pain. However, physical therapy requires active participation from patients in addition to lifestyle modifications. Additionally, for some patients, the severity of their musculoskeletal pain precludes them from effectively participating in physical therapy. For those patients, trigger point injections may provide enough relief to effectively participate in physical therapy. Trigger point injections is a procedure where an area identified is first injected with a local anesthetic then the needle is repeatedly inserted in and out (needling). The exact mechanism of action is not clear, but it does provide significant relief for most patients with musculoskeletal pain. Interestingly enough, while trigger point injections are a very common procedure and are performed by almost all pain physicians, there is great variability in the method it is performed. There is currently no clear guidance as to how light or intense the "needling" aspect of the procedure should be. On one end of the spectrum, some pain physicians perform 1-2 needle passes. On the opposite end of the spectrum, other pain physicians perform 40-50 or more needle passes. The literature is not very clear as to which is better in terms of the number of passes. In fact, the range of passes from one study to the other may account for some inconsistencies of the outcome associated with performing trigger point injections. The greater the number of passes, the greater the risk for possible side effects. On the other hand, pain relief may be directly proportional to the number of passes. The investigators currently do not have such information. The purpose of this study is to understand the relationship between the intensity of the needling aspect of trigger point injections and pain relief. In this study, patients will undergo the typical standard of care treatment for musculoskeletal pain with randomization regarding the number of passes during needling. The investigators will evaluate the patient response using paper surveys over 2 months following their procedures.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak, read and write English
* Diagnosis of myofascial pain
* Failed conservative therapy or unable to participate in physical therapy

Exclusion Criteria:

* Serious mental illness that may not enable the patient to perceive pain changes
* History of conditions which may present as diffuse pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2026-12-09 (Estimated); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | 60 days
  The primary outcome is the length of time patients subjectively report at least 50 percent reduction in pain compared to their baseline following trigger point injections using the Numerical Pain Scale which ranges from 0-10, where 0 = no pain and 10 = the worst possible pain.

SECONDARY OUTCOMES:
Change in Sleep patterns | 60 days
  Change the Pittsburgh Sleep Quality Assessment Questionnaire by at least 30 percent. The Pittsburgh Sleep Quality Assessment Questionnaire has a scale from 0-21. The lower the score, the better the sleep quality.
Perceived Subjective Changes in the Ability to Work, Do Chores, and Exercise. | 60 days
  Changes in abilities of the participants to work, do chores, and exercise by at least 30 percent. This will be assessed using subjective reports from the recruited participants. The participants will be asked to report their perceived changes in their ability to Work, do chores, and exercise. Zero percent indicates no change from baseline. one hundred percent indicates complete resolution of the perceived problem.

CONTACTS AND LOCATIONS:
Overall Officials: Mohab Ibrahim, Md., Ph.D, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center Multispecialty Services Clinic, Tucson, Arizona, United States